CLINICAL TRIAL: NCT04915716
Title: Effect of Fasting Time Before Cesarean Section on Neonatal Blood Glucose in Pregnant Women With Gestational Diabetes Mellitus
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: SAHoWMU-CR2021-07-202
Record Dates: First submitted 2021-06-04; First posted 2021-06-07 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: Gestational Diabetes Mellitus
Keywords: gestational diabetes mellitus; cesarean section; preoperative fasting; neonatal blood glucose
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- healthy pregnant woman: healthy pregnant woman
  Interventions: Other: Peripheral blood glucose levels were monitored
- pregnant women with GDM: pregnant women with gestational diabetes mellitus
  Interventions: Other: Peripheral blood glucose levels were monitored

INTERVENTIONS:
Other: Peripheral blood glucose levels were monitored — Peripheral blood glucose levels were monitored

SUMMARY:
Objective: To observe the effect of different fasting time on neonatal blood glucose in pregnant women with gestational diabetes mellitus (GDM). Methods: 122 pregnant women with gestational diabetes mellitus were selected from September 2018 to September 2020 in XX Hospital for regular prenatal examination, matching of pregnancy and delivery times, and undergoing elective lower uterine cesarean section to terminate pregnancy. The pregnant women were divided into 5 groups according to their fasting time before operation and whether they were given rehydration on the same day before operation, There were 27 cases in group B (fasting time 12.75 ± 0.48 hours, no rehydration before operation), 20 cases in group C (fasting time 15.65 ± 0.52 hours, no rehydration before operation), 24 cases in group D (fasting time 12.75 ± 0.48 hours, intravenous drip of 5% glucose sodium chloride 500ml at 8:00 on the day of operation), 24 cases in Group E (fasting time 15.65 ± 0.52 hours, intravenous drip of 5% glucose sodium chloride 500ml at 8:00 on the day of operation). The blood glucose of pregnant women within half an hour before operation, the blood glucose of newborns after delivery and the incidence of neonatal hypoglycemia were observed and recorded.

ELIGIBILITY:
Inclusion Criteria:

(1) The pregnant woman is born at term and has a single child; (2) Regular obstetric examination during pregnancy with complete obstetric examination data was diagnosed as gestational diabetes mellitus; (3) Pregnant women with body mass index (BMI) < 35kg/㎡; (4) All the operations were performed electively, and epidural anesthesia was used as the surgical anesthesia.

Exclusion Criteria:

(1) Pregnancy complicated with medical and surgical diseases, such as thyroid dysfunction and chronic hypertension; (2) Insufficiency of vital organ function or complicated tumor; (3) Pregnant women with other pregnancy complications besides GDM, such as preeclampsia, etc.; (4) The operation method is classical cesarean section or pregnant women with postpartum hemorrhage;

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
blood glucose concentration | 37 weeks to 40 weeks gestation
  Peripheral blood glucose concentration of maternal fingers

SECONDARY OUTCOMES:
blood glucose concentration | 37 weeks to 40 weeks gestation
  Blood glucose concentration in the peripheral finger of the newborn

IPD SHARING:
Plan to Share IPD: Undecided